CLINICAL TRIAL: NCT04842578
Title: The Guidance of Thin Cross- Section of CT in Anatomic Segmentectomy With or Without 3-dimensional Computed Tomography Lung Simulation
Brief Title: The Guidance of Thin Cross- Section of CT in Anatomic Segmentectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: thin cross- section of CT ZYP
Record Dates: First submitted 2021-04-03; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Segmentectomy; Video- Assisted Thoracoscopic Surgery; Three-dimensional-computed Tomography (3D-CT); Thin Cross- Section of CT

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group of thin cross- section of CT (Experimental): Anatomic Segmentectomy with the Guidance of Thin Cross- Section of CT
  Interventions: Other: Cross- Section of CT Guided Anatomic Segmentectomy
- group of thin 3D simulation (Active Comparator): Anatomic Segmentectomy with the Guidance of 3D simulation
  Interventions: Other: 3D simulation Guided Anatomic Segmentectomy

INTERVENTIONS:
Other: Cross- Section of CT Guided Anatomic Segmentectomy — The anatomic segmentectomy is base on the reading and comprehension of Cross- Section of CT.
  Arms: group of thin cross- section of CT
Other: 3D simulation Guided Anatomic Segmentectomy — The anatomic segmentectomy is base on the overview of 3D simulation of pulmonary structure.
  Arms: group of thin 3D simulation

SUMMARY:
Three-dimensional (3D) simulation of pulmonary vessels and the space between the lesion and adjacent tissues is regarded improving the safety and accuracy of video-assisted thoracoscopic surgery (VATS) for segmentectomy for ground glass opacity (GGO) in lung. However, not every thoracic surgeon can handle the technique, in addition, the 3D reconstruction originate from the thin CT scan. Actually, the investigators found that, the reading and comprehension of the thin cross- section of CT can guide the accurate anatomic segmentectomy in most situations. The investigators designed a retrospective study to compare the reading of thin cross- section of CT with 3D reconstruction or without 3D reconstruction during the guidance of anatomic segmentectomy.

ELIGIBILITY:
Inclusion Criteria:

Selection criteria for VATS segmentectomy in the present study were as follows:

(I) patients with single peripheral GGO lesion considered suspicious for malignancy;

(II) the lesion <2 cm in diameter and with at least one of the followings:

(i) pure adenocarcinoma in situ (AIS) histology;

(ii) nodule has ≥50% ground-glass appearance on high resolution CT;

(iii) radiologic surveillance conforms a long doubling time (≥400 days).

Exclusion Criteria:

(I) patients with insufficient cardiopulmonary function;

(II) other contraindication for segmentectomy.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
planning time (minutes) | from the first time of thin cross- section of CT is presented to the end of surgery, within 7 days
  the planning time for anatomic segmentectomy before surgery, including the time- cost of the decision making and the planning time for surgery
time before surgery (days) | from the day of being hospitalized to the day of surgery, within 5 days
  days before surgery after being hospitalized
operation time (minutes) | from beginning to the end of surgery, up to 180 minutes
  the duration of the operation time
confirmation time during surgery （number） | Intraoperative
  review time of the 3D reconstruction or the thin cross- section of CT during surgery
air leakage after surgery (days) | within 7 days after surgery
  the days of air leakage after surgery
the incidence of pneumonia （percentage） | within 7 days after surgery
  the incidence of pneumonia after surgery
the incidence of atelectasis （percentage） | within 7 days after surgery
  the incidence of atelectasis after surgery
Intraoperative bleeding (ml) | Intraoperative
  bleeding during anatomic segmentectomy, through the operation, an average of 100 ml
Chest tube duration (days) | within 7 days after surgery
  Chest tube duration after surgery
Postoperative hospital stay (days) | within 7 days after surgery
  hospital stay after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xiaogang Zhao, Study Director — The Second Hospital of Shandong University
Locations (1):
- The Second Hospital of Shandong University, Jinan, Shandong, China